CLINICAL TRIAL: NCT03246087
Title: Acupuncture for Plantar Fasciosis in the Primary Care Setting
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mike O'Callaghan Military Hospital (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: FWH20170077H
Record Dates: First submitted 2017-07-14; First posted 2017-08-11 (Actual); Results first posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Plantar Fascitis
Keywords: acupuncture; plantar fasiosis
MeSH Terms: interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Acupuncture (Active Comparator): Patients will receive acupuncture for plantar fasciosis. The standard of care home exercise program will be reviewed along with the stretching and strengthening exercises.
  Interventions: Device: Acupunture
- Standard of Care (Experimental): The standard of care home exercise program will be reviewed along with the stretching and strengthening exercises.
  Interventions: Other: Standard of care
- Crossover (Experimental): At the end of the study, patients in the Standard of Care group whom are still experiencing pain and symptoms will be rolled into the acupuncture treatment arm of the study.
  Interventions: Device: Acupunture

INTERVENTIONS:
Device: Acupunture — acupuncture for plantar fasciosis
  Acupuncture will be performed and the standard of care prescribed home exercise program will be reviewed.
  Arms: Acupuncture; Crossover
Other: Standard of care — standard of care home exercise program
  Arms: Standard of Care

SUMMARY:
The purpose of this study is to determine if the addition of acupuncture to a standard of care prescribed exercise program is more effective at improving pain and function in adult patients with plantar fasciosis.

DETAILED DESCRIPTION:
Investigators are studying whether a specific acupuncture protocol, when added to the standard of care treatment, can improve pain and function in adults with plantar fasciosis. Investigators hypothesize that there will be a significant improvement in both pain and functional outcomes, both acutely and over time, in the experimental group compared to the control group. Investigators will measure foot pain immediately prior to treatment (baseline), immediately after the initial treatment and at 2 weeks, 4 weeks, and 3 months. The Foot Function Index Revised short form will be used during the same intervals to evaluate foot function. At 3 months, patients in the non-acupuncture group will cross-over into the acupuncture group if still experiencing pain.

ELIGIBILITY:
THIS STUDY IS BEING CONDUCTED AT A MILITARY INSTALLATION. YOU MUST HAVE MILITARY INSURANCE IN ORDER TO PARTICIPATE IN THIS STUDY.

Inclusion Criteria:

Male and female DoD beneficiaries, age 18 years or older, who have been diagnosed with plantar fasciitis/fasciosis OR Patients meeting criteria of pain in the bottom of the foot/heel with first steps in the morning & tender to palpation over the medial calcaneal tubercle (where the plantar fascia inserts). Those with acute and chronic diagnoses will be included.

Exclusion Criteria:

* Pregnant
* Absence of leg
* Active cellulitis of lower extremity
* Prior surgery for plantar fasciitis
* Steroid injections in the last 12 weeks for plantar fasciitis; if received in last 12 weeks subjects will be offered to be involved in the study after they have completed a 12 week wash out period.
* Any regenerative therapy to include proliferation therapy or platelet rich plasma therapy in the last 12 weeks for plantar fasciitis; if received in last 12 weeks subject will be offered to be involved in the study after they have completed a 12 week wash out period.
* Botox injections for plantar fasciitis injections in the last 12 weeks for plantar fasciitis; if received in last 12 weeks subject will be offered to be involved in the study after they have completed a 12 week wash out period.
* Use of anticoagulants
* If they have every had any prior acupuncture for plantar fasciitis using the defined KB-2 points

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Actual)
Dates: Start 2017-10-17 (Actual); Primary Completion 2019-04-13 (Actual); Study Completion 2019-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Cagle, MD, Principal Investigator — Scott AFB; Carlton Covey, MD, Principal Investigator — Nellis AF
Locations (2):
- United States (2):
  - Scott AFB, Belleville, Illinois
  - Mike O'Callaghan Federal Hospital, Nellis Air Force Base, Nevada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cotchett MP, Landorf KB, Munteanu SE. Effectiveness of dry needling and injections of myofascial trigger points associated with plantar heel pain: a systematic review. J Foot Ankle Res. 2010 Sep 1;3:18. doi: 10.1186/1757-1146-3-18. PMID 20807448
- [Background] Covey CJ, Mulder MD. Plantar fasciitis: How best to treat? J Fam Pract. 2013 Sep;62(9):466-71. PMID 24080555
- [Background] Glickman-Simon R, Wallace J. Acupuncture for knee osteoarthritis, chasteberry for premenstrual syndrome, probiotics for irritable bowel syndrome, yoga for hypertension, and trigger point dry needling for plantar fasciitis. Explore (NY). 2015 Mar-Apr;11(2):157-61. doi: 10.1016/j.explore.2014.12.009. Epub 2014 Dec 29. No abstract available. PMID 25682385
- [Background] Kumnerddee W, Pattapong N. Efficacy of electro-acupuncture in chronic plantar fasciitis: a randomized controlled trial. Am J Chin Med. 2012;40(6):1167-76. doi: 10.1142/S0192415X12500863. PMID 23227789
- [Background] Li S, Shen T, Liang Y, Zhang Y, Bai B. Miniscalpel-Needle versus Steroid Injection for Plantar Fasciitis: A Randomized Controlled Trial with a 12-Month Follow-Up. Evid Based Complement Alternat Med. 2014;2014:164714. doi: 10.1155/2014/164714. Epub 2014 Jul 8. PMID 25114704
- [Background] Schwartz O, Levinson T, Astman N, Haim L. Attrition due to orthopedic reasons during combat training: rates, types of injuries, and comparison between infantry and noninfantry units. Mil Med. 2014 Aug;179(8):897-900. doi: 10.7205/MILMED-D-13-00567. PMID 25102533
- [Background] Owens BD, Wolf JM, Seelig AD, Jacobson IG, Boyko EJ, Smith B, Ryan MA, Gackstetter GD, Smith TC; Millennium Cohort Study Team. Risk Factors for Lower Extremity Tendinopathies in Military Personnel. Orthop J Sports Med. 2013 Jun 11;1(1):2325967113492707. doi: 10.1177/2325967113492707. eCollection 2013 Jan-Jun. PMID 26535232
- [Background] Roy TC. Diagnoses and mechanisms of musculoskeletal injuries in an infantry brigade combat team deployed to Afghanistan evaluated by the brigade physical therapist. Mil Med. 2011 Aug;176(8):903-8. doi: 10.7205/milmed-d-11-00006. PMID 21882780
- [Background] Scher DL, Belmont PJ Jr, Bear R, Mountcastle SB, Orr JD, Owens BD. The incidence of plantar fasciitis in the United States military. J Bone Joint Surg Am. 2009 Dec;91(12):2867-72. doi: 10.2106/JBJS.I.00257. PMID 19952249
- [Background] Thiagarajah AG. How effective is acupuncture for reducing pain due to plantar fasciitis? Singapore Med J. 2017 Feb;58(2):92-97. doi: 10.11622/smedj.2016143. Epub 2016 Aug 16. PMID 27526703
- [Background] Woitzik E, Jacobs C, Wong JJ, Cote P, Shearer HM, Randhawa K, Sutton D, Southerst D, Varatharajan S, Brison RJ, Yu H, van der Velde G, Stern PJ, Taylor-Vaisey A, Stupar M, Mior S, Carroll LJ. The effectiveness of exercise on recovery and clinical outcomes of soft tissue injuries of the leg, ankle, and foot: A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Man Ther. 2015 Oct;20(5):633-45. doi: 10.1016/j.math.2015.03.012. Epub 2015 Mar 28. PMID 25892707
- [Background] Zhang SP, Yip TP, Li QS. Acupuncture treatment for plantar fasciitis: a randomized controlled trial with six months follow-up. Evid Based Complement Alternat Med. 2011;2011:154108. doi: 10.1093/ecam/nep186. Epub 2011 Feb 15. PMID 19933769

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 94 total subjects. 78 total subjects analyzed. 39 from the initial placebo group were allowed to crossover once their placebo study role was completed.
Groups:
- Acupuncture: Patients will receive acupuncture for plantar fasciosis. The standard of care home exercise program will be reviewed along with the stretching and strengthening exercises.
  Acupunture: acupuncture for plantar fasciosis
  Acupuncture will be performed and the standard of care prescribed home exercise program will be reviewed.
- Crossover: At the end of the study, patients in the Standard of Care group whom are still experiencing pain and symptoms will be rolled into the acupuncture treatment arm of the study.
  Acupunture: acupuncture for plantar fasciosis
  Acupuncture will be performed and the standard of care prescribed home exercise program will be reviewed.
Period: Randomized
Arm/Group | Acupuncture | Standard of Care | Crossover
Started | 47 | 47 | 0
Completed | 39 | 39 | 0
Not Completed | 8 | 8 | 0
Period: Crossover to Acupuncture
Arm/Group | Acupuncture | Standard of Care | Crossover
Started | 0 | 0 | 39
Completed | 0 | 0 | 30
Not Completed | 0 | 0 | 9

BASELINE CHARACTERISTICS:
Population: 39 of the 47 Standard of care crossed over.
Groups:
- Total: Total of all reporting groups
Arm/Group | Acupuncture | Standard of Care | Crossover | Total
Number analyzed (Participants) | 47 | 47 | 0 | 94
Age, Customized [Mean (Standard Deviation); unit: years]
  age | 41 (12) | 45 (12) |  | 43 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 25 | 24 | 0 | 49
  Male | 22 | 23 | 0 | 45
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 6 | 0 | 10
  Not Hispanic or Latino | 43 | 41 | 0 | 84
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 2 | 0 | 0 | 2
  Asian | 3 | 2 | 0 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 10 | 12 | 0 | 22
  White | 27 | 25 | 0 | 52
  More than one race | 5 | 8 | 0 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 47 | 47 |  | 94
foot injury history [Number; unit: participants]
  foot injury history-yes | 36 | 32 |  | 68
  foot injury history-no | 11 | 15 |  | 26

OUTCOME MEASURES:

1. Primary Outcome: NPRS-11
Description: Numeric Pain Rating Scale. 11 point numeric rating on a scale of 0-10 to measure pain intensity. 0 being no pain, 5 being moderate pain, and 10 being worst pain.
Time Frame: 90 days
Population: Crossover pulls from the standard of care group. There are not 30 additional subjects, merely 30 subjects pulled from standard of care to crossover to acupuncture group.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Standard of Care | Crossover
Number analyzed (Participants) | 39 | 39 | 30
score on a scale
  week 0 | 3.8 (2.4) | 4.3 (2.8) | 3.7 (2.7)
  week 2 | 3.1 (2.3) | 3.7 (2.8) | 3.0 (2.6)
  week 4 | 2.6 (2.1) | 3.3 (2.5) | 2.1 (2.0)
  week 6 | 2.5 (2.2) | 3.0 (2.2) | 2.6 (2.2)
  week 12 | 2.4 (2.2) | 3.4 (2.8) | 2.6 (2.2)

2. Secondary Outcome: FFI-R
Description: Revised Foot Function Index Short Form. FFI-R measures the impact of foot pathology on function for 5 subscales of: pain (7 questions), stiffness (7 questions), difficulty (11 questions), activity limitation (3 questions), social issues (6 questions).
  Each question ranges from 1 (no pain/no stiffness/no difficulty/none of the time) to 4 (severe pain/stiffness/difficulty/all of the time).
  Subscale scores are added up to a total cumulative score. Minimum total score (least pain/stiffness/difficulty) is 34. Maximum total score (most pain/stiffness/difficulty) is 136.
Time Frame: 90 days
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Acupuncture | Standard of Care | Crossover
Number analyzed (Participants) | 39 | 39 | 39
score on a scale
  week 0: number analyzed (Participants) | 39 | 39 | 37
  week 0 | 73 (14) | 70 (22) | 63 (17)
  week 2 | 61 (16) | 64 (23) | 60 (22)
  week 4 | 56 (16) | 60 (21) | 55 (22)
  week 6 | 56 (18) | 58 (21) | 58 (23)
  week 12 | 52 (18) | 55 (21) | 56 (24)

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Acupuncture | Standard of Care | Crossover
All-Cause Mortality (participants affected / at risk) | 0/47 | 0/47 | 0/39
Serious Adverse Events (participants affected / at risk) | 0/47 | 0/47 | 0/39
Other Adverse Events (participants affected / at risk) | 4/47 | 1/47 | 0/39
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Acupuncture (N=47) | Standard of Care (N=47) | Crossover (N=39)
Non Serious Adverse Event (Musculoskeletal and connective tissue disorders) | 4 (4) | 0 (0) | 0 (0)
Non Serious Adverse Event (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-24): https://cdn.clinicaltrials.gov/large-docs/87/NCT03246087/Prot_SAP_000.pdf